CLINICAL TRIAL: NCT06301685
Title: Effectiveness of Lidocaine Injection on Stellate Ganglion in Pediatric Patients With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Effectiveness of Lidocaine Injection on Stellate Ganglion in Pediatric Patients With Autism Spectrum Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-AST
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Injections; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine therapy+Stellate ganglion block (Experimental): The study lasts 10 days for each patient. During the treatment, All the participants are provided with the routine rehabilitation therapy.
  Based on the invention above, the patients were provided with stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g)
  Interventions: Behavioral: Routine therapy; Procedure: Injection; Drug: Lidocaine Hydrochloride
- Routine therapy+Placebo (Placebo Comparator): The study lasts 20d for each patient. During the treatment, All the participants are provided with the routine rehabilitation therapy and placebo injection.
  Interventions: Behavioral: Routine therapy; Procedure: Injection

INTERVENTIONS:
Behavioral: Routine therapy — The study lasts 10 days for each patient. During the treatment, All the participants are provided with the routine therapy, which included routine rehabilitation, cognitive training.
Procedure: Injection — The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
Drug: Lidocaine Hydrochloride — the patients were provided with Stellate ganglion block , using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck. once a day.
  Other Names: Lidocaine
  Arms: Routine therapy+Stellate ganglion block

SUMMARY:
The goal of this clinical trial is to explore efficacy of stellate ganglion block Children with Autistic Disorder. The main question it aims to answer is:

Can stellate ganglion block improve the Autistic Disorder in children? Children with Autistic Disorder will be divided into the control group and experimental group evenly. All the patients were provided with routine therapy, while the patients in the experimental group were given stellate ganglion block. The Childhood Autism Rating Scale of the two groups of patients before and after treatment are evaluated.

DETAILED DESCRIPTION:
Autistic Disorder in children is becoming increasingly more. The goal of this clinical trial is to explore efficacy of stellate ganglion block Children with Autistic Disorder. The main question it aims to answer is:

Can stellate ganglion block improve the Autistic Disorder in children? Children with Autistic Disorder will be divided into the control group and experimental group evenly. All the patients were provided with routine therapy, while the patients in the experimental group were given stellate ganglion block. The Childhood Autism Rating Scale of the two groups of patients before and after treatment are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Autistic Disorder.
* Aged between 3 years old and 6 years old.
* No contraindications to stellate ganglion block.

Exclusion Criteria:

* Other significant physical or neurodevelopmental disorders.
* Other significant medical conditions

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale | day 1 and day 10
  In the Childhood Autism Rating Scale, the rater observes the behavior of the child in specific situations and assigns scores based on a series of descriptive items. Each item is scored on a range of 0 to 4, with 0 indicating no abnormality and 4 indicating severe abnormality. The rater also considers the overall impression and severity of the child, resulting in a total score. The total score falls between 15 and 60, with higher scores indicating a higher level of autism severity.

SECONDARY OUTCOMES:
Children's Communication Checklist | day 1 and day 10
  This checklist was to assess language abilities in children aged 2-16. It consists of 70 items divided into eight subscales, including vocabulary, grammar, comprehension, expression, communication, regulation, fluency, and nonverbal communication. Scores range from 0-280, with higher scores indicating better language ability.
Social Interaction Assessment Scale | day 1 and day 10
  This scale was developed by American psychiatrist Eric Schopler and colleagues to assess social interaction and behavior in children with autism and related disorders. It consists of 29 items divided into three subscales, including social interaction, maladaptive behavior, and language/communication. Scores range from 0-87, with higher scores indicating better social interaction and behavior.
Children's Depression Inventory | day 1 and day 10
  This inventory was developed by American psychologist Maria Kovacs to assess depression in children aged 7-17. It consists of 27 items covering aspects such as sad mood, self-evaluation, life satisfaction, insomnia, and early morning awakening. Scores range from 0-54, with higher scores indicating greater severity of depression.
Childhood Anxiety Sensitivity Index | day 1 and day 10
  This index was developed by Australian psychologist Ronald Rapee and colleagues to assess anxiety sensitivity in children aged 8-15. It consists of 18 items covering physical sensations, cognition, and behavior. Scores range from 0-54, with higher scores indicating greater anxiety sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group

IPD SHARING:
Plan to Share IPD: No